CLINICAL TRIAL: NCT02577029
Title: A Multicenter, Open-Label Study to Evaluate ARC-520 Administered Alone and in Combination With Other Therapeutics in Patients With Chronic Hepatitis B Virus (HBV) Infection (MONARCH)
Brief Title: Study of ARC-520 With or Without Other Drugs Used in the Treatment of Chronic Chronic Hepatitis B Virus (HBV)
Acronym: MONARCH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heparc-2008; 2015-005499-46 (EudraCT Number)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B; Hepatitis D
MeSH Terms: conditions — Hepatitis B; Hepatitis D | interventions — ARC-520; entecavir; peginterferon alfa-2a; Tenofovir; Histamine Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (Experimental): Treatment-naïve, hepatitis B "e" antigen (HBeAg)-positive participants with chronic hepatitis B (CHB) of any genotype administered ARC-520 (2 mg/kg intravenous [IV]) every 4 weeks for 48 weeks (13 doses).
  Interventions: Drug: ARC-520; Drug: antihistamine
- Cohort 2 (Experimental): Treatment-naïve, HBeAg-positive, Genotype B participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered ETV or TDF for approximately 60 weeks starting Day 1 and weekly subcutaneously administered peginterferon (PEG IFN) alpha 2a for 48 weeks starting Day 87.
  Interventions: Drug: ARC-520; Drug: entecavir; Biological: pegylated interferon alpha 2a; Drug: tenofovir disoproxil; Drug: antihistamine
- Cohort 3 (Experimental): Treatment-naïve, HBeAg-negative, Genotype B participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered ETV or TDF for approximately 60 weeks starting Day 1 and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 87.
  Interventions: Drug: ARC-520; Drug: entecavir; Biological: pegylated interferon alpha 2a; Drug: tenofovir disoproxil; Drug: antihistamine
- Cohort 4 (Experimental): Treatment-naïve, HBeAg-positive, Genotype C participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered ETV or TDF for approximately 60 weeks starting Day 1 and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 87.
  Interventions: Drug: ARC-520; Drug: entecavir; Biological: pegylated interferon alpha 2a; Drug: tenofovir disoproxil; Drug: antihistamine
- Cohort 5 (Experimental): Treatment-naïve, HBeAg-negative, Genotype C participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered ETV or TDF for approximately 60 weeks starting Day 1 and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 87.
  Interventions: Drug: ARC-520; Drug: entecavir; Biological: pegylated interferon alpha 2a; Drug: tenofovir disoproxil; Drug: antihistamine
- Cohort 6 (Experimental): Treatment-naïve, HBeAg-negative, Genotype D participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered ETV or TDF for approximately 60 weeks starting Day 1 and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 87.
  Interventions: Drug: ARC-520; Drug: entecavir; Biological: pegylated interferon alpha 2a; Drug: tenofovir disoproxil; Drug: antihistamine
- Cohort 7 (Experimental): Treatment-naïve, HBeAg-negative or HBeAg-positive participants with hepatitis delta virus (HDV) administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 15.
  Interventions: Drug: ARC-520; Biological: pegylated interferon alpha 2a; Drug: antihistamine
- Cohort 8 (Experimental): Treatment-naïve, HBeAg-positive participants with CHB of any genotype administered ARC-520 (4 mg/kg IV) every 4 weeks for 48 weeks (13 doses).
  Interventions: Drug: ARC-520; Drug: antihistamine

INTERVENTIONS:
Drug: ARC-520 — ARC-520 will be administered intravenously concomitantly with 0.9% normal saline using an infusion rate of 0.4 mL/min (24 mL/hour) for study treatment and 200 mL/hr for saline.
Drug: entecavir — 0.5 mg once daily; oral
  Other Names: Baraclude
  Arms: Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6
Biological: pegylated interferon alpha 2a — 180 mcg; subcutaneous injection once weekly
  Other Names: Peginterferon; Pegasys
  Arms: Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7
Drug: tenofovir disoproxil — 300 mg once daily; oral
  Other Names: Viread
  Arms: Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6
Drug: antihistamine — All participants will be pre-treated with an oral antihistamine selected by the investigator from the list of approved antihistamines that is available in that country. Acceptable antihistamines are: diphenhydramine 50 mg p.o., chlorpheniramine 8 mg p.o., hydroxyzine 50 mg p.o., or cetirizine 10 mg p.o.

SUMMARY:
Patients with chronic HBV infection will receive either ARC-520 alone or ARC-520 in combination with other treatments such as entecavir (ENT) or tenofovir (TDF) and/or pegylated interferon (PEG IFN) alpha 2a therapy, and be evaluated for safety and efficacy.

DETAILED DESCRIPTION:
This is a multicenter, open-label study of ARC-520 based treatment regimens administered to patients with HBeAg positive or HBeAg negative immune active chronic Hepatitis B Virus (HBV) infection of various genotypes, or patients with Hepatitis D Virus (HDV). Eligible patients naive to previous treatment, and who have signed an Ethics Committee - approved informed consent, will be enrolled and will receive ARC-520 alone or ARC-520 plus additional treatments such as entecavir (ETV) or tenofovir (TDF) and/or pegylated interferon alpha 2a (PEG IFN) therapy. The study may initially involve up to a total of 96 eligible chronic HBV and HDV infected patients. Patients in all cohorts will receive a total of 13 doses of ARC-520 at 2mg/kg or 4 mg/kg. Patients will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate, and temperature), weight, adverse events assessment (AEs), 12-lead ECGs, liver fibrosis testing, concomitant medication assessment, blood sample collection for hematology, coagulation, chemistry, exploratory Pharmacodynamic (PD) measures, urinalysis, HBV serology, cytokines, Follicle Stimulating Hormone (FSH) testing (post-menopausal females) and pregnancy testing for females of childbearing potential. Clinically significant changes including AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the patient is lost to follow-up. For each patient, the duration of the study is approximately 96 weeks, from enrolment to last visit. Prior to enrolment there is a 60 day screening period. Addition of new cohorts and additional treatment regimens are anticipated for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Written informed consent
* No clinically significant abnormalities at screening/pre-dose 12-lead ECG assessment
* Diagnosis of HBeAg negative or positive chronic HBV infection.
* Must be HBsAg (+) during screening.
* Must be treatment naïve: never on PEG IFN alpha 2a and/or ETV or TDF; and
* Have not used nucleoside/nucleotide analogs (NUCs) within the last 2 years prior to dosing on Day 1
* Must use 2 effective methods of contraception (double barrier contraception or hormonal contraceptive along with a barrier contraceptive) (both male and female partners)

Exclusion Criteria:

* Pregnant or lactating
* Acute signs of hepatitis/other severe infections within 4 weeks of screening
* Use within the last 14 days or anticipated requirement for anticoagulants, systemic corticosteroids, immunomodulators, or immunosuppressants
* Use of prescription medication within 14 days prior to treatment administration except: topical products without systemic absorption, statins (except rosuvastatin), hypertension medications, over-the-counter (OTC) and prescription pain medication or hormonal contraceptives
* History of poorly controlled autoimmune disease or any history of autoimmune hepatitis
* History of heterozygous or homozygous familial hypercholesterolemia.
* Human immunodeficiency virus (HIV) infection
* Is sero-positive for Hepatitis C Virus (HCV), or has a history of delta virus hepatitis (except for cohort in which delta virus infection is acceptable)
* Has hypertension: blood pressure > 170/100 mmHg; well-controlled blood pressure on hypertensive medication allowed
* History of cardiac rhythm disturbances
* Family history of congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease within 6 months prior to study entry
* History of malignancy, except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer
* Has had major surgery within 1 month of screening
* Regular use of alcohol within 6 months prior to screening (ie, more than 14 units of alcohol per week)
* Use of recreational drugs such as cocaine, phencyclidine (PCP), and methamphetamines, within 1 year prior to the screening
* History of allergy to bee sting
* Clinically significant history of any alcoholic liver disease, cirrhosis, Wilson's disease, hemochromatosis, or alpha-1 antitrypsin deficiency
* Presence of cholangitis, cholecystitis, cholestasis, or duct obstruction
* Clinically significant history or presence of poorly controlled/uncontrolled systemic disease
* Presence of any medical or psychiatric condition or social situation that impacts compliance or results in additional safety risk
* History of coagulopathy/stroke within past 6 months, and/or concurrent anticoagulant medication(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- Australia (9):
  - Research Site 3, Camperdown, New South Wales
  - Research Site 8, Concord, New South Wales
  - Research Site 5, Darlinghurst, New South Wales
  - Research Site 1, Westmead, New South Wales
  - Research Site 9, Adelaide, South Australia
  - Research Site 6, Clayton, Victoria
  - Research Site 4, Fitzroy, Victoria
  - Research Site 2, Parkville, Victoria
  - Research Site 7, Nedlands, Washington
- Bulgaria (4):
  - Research Site 13, Pleven
  - Research Site 10, Sofia
  - Research Site 11, Sofia
  - Research Site 12, Varna
- Research Site 14, Hong Kong, China
- Research Site 25, Chisinau, Moldova
- New Zealand (3):
  - Research Site 23, Papatoetoe, Aukland
  - Research Site 24, Dunedin, Otago-Southland
  - Research Site 21, Auckland
- South Korea (6):
  - Research Site 17, Busan
  - Research Site 19, Busan
  - Research Site 16, Daegu
  - Research Site 18, Seoul
  - Research Site 15, Seoul
  - Research Site 20, Seoul
- Taiwan (3):
  - Research Site 27, Douliu, Yunlin County
  - Research Site 26, Changhua
  - Research Site 28, Kaohsiung City
- Thailand (6):
  - Research Site 29, Bangkok
  - Research Site 30, Bangkok
  - Research Site 32, Bangkok
  - Research Site 33, Chiang Mai
  - Research Site 31, Khon Kaen
  - Research Site 34, Pathum Thani

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: Treatment-naïve, HBeAg-positive, Genotype B participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered entecavir (ETV) or tenofovir (TDF) for approximately 60 weeks starting Day 1 and weekly subcutaneously administered peginterferon (PEG IFN) alpha 2a for 48 weeks starting Day 87.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Started | 10 | 2 | 7 | 12 | 11 | 13 | 12 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 2 | 7 | 12 | 11 | 13 | 12 | 12
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Termination of the Study | 9 | 2 | 5 | 12 | 10 | 12 | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Treatment-naïve, HBeAg-positive participants with CHB of any genotype administered ARC-520 (2 mg/kg IV) every 4 weeks for 48 weeks (13 doses).
- Cohort 2: Treatment-naïve, HBeAg-positive, Genotype B participants with CHB administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) concomitantly with daily orally administered ETV or TDF for approximately 60 weeks starting Day 1 and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 87.
- Cohort 7: Treatment-naïve, HBeAg-negative or HBeAg-positive participants with HDV administered ARC-520 (2 mg/kg increasing to 4 mg/kg or 4 mg/kg IV) every 4 weeks for 48 weeks (13 doses) and weekly subcutaneously administered PEG IFN alpha 2a for 48 weeks starting Day 15.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Total
Number analyzed (Participants) | 10 | 2 | 7 | 12 | 11 | 13 | 12 | 12 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (11.09) | 29.5 (0.71) | 40.4 (7.37) | 36.3 (9.32) | 39.6 (12.61) | 38.2 (7.97) | 39.6 (7.73) | 36.7 (7.32) | 37.4 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 4 | 6 | 3 | 2 | 6 | 5 | 34
  Male | 3 | 1 | 3 | 6 | 8 | 11 | 6 | 7 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 1-log Reduction in Hepatitis B Surface Antigen (HBsAg) at Week 60 Compared to Baseline
Description: The percentage of participants with chronic HBV achieving a 1-log reduction in HBsAg compared to baseline (mean of pre-dose values) at Week 60 after completion of 48 weeks of ARC-520 Injection.
Time Frame: Baseline, Week 60
Population: The study was terminated prior to any participant reaching Week 60 of treatment; therefore, this outcome measure could not be analyzed.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs Considered Possibly or Probably Related to Treatment
Description: The Principal Investigator (or medically qualified designee) will use clinical judgment to determine the relationship. An adverse event (AE) was considered "possibly related" when there is a reasonable possibility that the incident, experience, or outcome may have been caused by the product under investigation. An AE was considered "probably related" when there are facts, evidence, or arguments to suggest that the event is related to the product under investigation. Only AEs that occurred post-dose were considered treatment-emergent. Clinically significant abnormal laboratory findings or other abnormal assessments that are detected during the study or are present at baseline and significantly worsen following the start of the study will be reported as AEs.
Time Frame: From first dose of study drug up to 36 weeks of treatment, plus up to 48 weeks of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 10 | 2 | 7 | 12 | 11 | 13 | 12 | 12
Participants
  Related TEAE | 1 | 0 | 3 | 2 | 3 | 4 | 3 | 3
  Related Serious TEAE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Percentage of Participants With HBsAg Loss (Based on Qualitative Assay) Over Time
Description: The qualitative HBsAg assay gives a binary result, positive or negative.
Time Frame: Weeks 52, 60, 72 and 96
Population: The study was terminated prior to any participant reaching Week 52 of treatment; therefore, this outcome measure could not be analyzed.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving a 1-log Reduction in HBsAg and Achieving an HBsAg Level < 100 IU/L Over Time
Time Frame: Weeks 52, 60, 72 and 96
Population: as for outcome 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to HBsAg Loss
Time Frame: Baseline through Week 96
Population: This analysis was not done since no events of HBsAg loss were observed to to Week 36. (No participant reached Week 96 of treatment due to study termination).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Time to Anti-HBs (Antibody to Hepatitis B Surface Antigen) Seroconversion
Time Frame: Baseline through Week 96
Population: as for outcome 5
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Anti-HBs Seroconversion Over Time
Time Frame: Weeks 52, 60, 72 and 96
Population: as for outcome 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With HBeAg Loss and Anti-Hepatitis B e Antigen (Anti-HBe) Seroconversion (if HBeAg-Positive at Study Entry) Over Time
Time Frame: Weeks 52, 60, 72 and 96
Population: as for outcome 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Resistance to ARC-520 Injection by Week 52
Description: Resistance is defined as > 1.0 log IU/mL quantitative HBsAg (qHBsAg) increase from nadir, confirmed by repeat test.
Time Frame: Week 52
Population: as for outcome 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Resistance to the Combination Therapy From Baseline to Week 60
Description: Resistance is defined as > 1.0 log IU/mL increase in HBV DNA from nadir, confirmed by repeat test.
Time Frame: Baseline, Week 60
Population: as for outcome 1
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With HDV With Undetectable HDV Ribonucleic Acid (RNA) After 48 Weeks of Concomitant ARC-520 Injection and PEG IFN Alpha 2a Therapy Over Time (Cohort 7 Only)
Time Frame: Weeks 52, 60, 72 and 96
Population: as for outcome 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Log Change From Baseline in Quantitative HBV Deoxyribonucleic Acid (DNA) Serum Levels Over Time
Time Frame: Baseline, Weeks 52, 60, 72 and 96
Population: as for outcome 1
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 36 weeks of treatment, plus up to 48 weeks of follow-up
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/7 | 0/12 | 0/11 | 1/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/10 | 0/2 | 4/7 | 5/12 | 5/11 | 8/13 | 9/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=2) | Cohort 3 (N=7) | Cohort 4 (N=12) | Cohort 5 (N=11) | Cohort 6 (N=13) | Cohort 7 (N=12) | Cohort 8 (N=12)
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=2) | Cohort 3 (N=7) | Cohort 4 (N=12) | Cohort 5 (N=11) | Cohort 6 (N=13) | Cohort 7 (N=12) | Cohort 8 (N=12)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Administration site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 3 | 3 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hot flush (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Peripheral coldness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Somnolence (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hernia repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The ARC-520 Injection development program was terminated early for regulatory and business reasons secondary to findings occurring in a non-clinical toxicology study. Program termination was not due to safety findings in humans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No